CLINICAL TRIAL: NCT00425386
Title: A Dose Escalation Phase II Study of Sunitinib Plus Erlotinib in Advanced Renal Carcinoma
Brief Title: Sunitinib and Erlotinib in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Ryan, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000526204; P30CA069533 (NIH); OHSU-2683 (Other: Oregon Health & Science University IRB); OHSU-SOL-06051-LM (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Results first posted 2012-02-16 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; clear cell renal cell carcinoma; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Erlotinib Hydrochloride; Sunitinib; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib and Sunitinib (Experimental): Drug: erlotinib hydrochloride Dose Level 0 = 50 mg/day, continuous daily; 0.5= 75 mg/day, continuous daily;
  1. 100 mg/day, continuous daily; 1.5= 125 mg/day, continuous daily;
  2. 150 mg/day, continuous daily
  Drug: sunitinib malate Will be administered at 50 mg daily, 4 weeks on, 2 weeks off
  Interventions: Drug: erlotinib hydrochloride; Drug: sunitinib malate; Procedure: biopsy

INTERVENTIONS:
Drug: erlotinib hydrochloride — Dose Level 0 = 50 mg/day, continuous daily; 0.5= 75 mg/day, continuous daily;
  1. 100 mg/day, continuous daily; 1.5= 125 mg/day, continuous daily;
  2. 150 mg/day, continuous daily
Drug: sunitinib malate — Will be administered at 50 mg daily, 4 weeks on, 2 weeks off
Procedure: biopsy — Paraffin block (or unstained slides) of the primary tumor and/or metastatic lesions (as available) and a plasma sample for future correlative studies will be collected. A paraffin block (or at least 10 unstained slides, each of 10 micromillimeter thickness) from the original paraffin-embedded biopsy material taken at the diagnosis will be stored at 4 degrees Celsius.

SUMMARY:
RATIONALE: Sunitinib and erlotinib may stop the growth of tumor cell by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib together with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying the best dose of erlotinib when given together with sunitinib and to see how well they work in treating patients with unresectable or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of erlotinib hydrochloride when administered with sunitinib malate in patients with unresectable or metastatic renal cell carcinoma.
* Determine the 8-month progression-free survival of patients treated with this regimen.

Secondary

* Determine the safety of sunitinib malate and erlotinib hydrochloride in these patients.
* Determine the duration of response in these patients.
* Determine the proportion of patients whose best overall response is complete response, partial response, stable disease, or progressive disease.
* Determine the overall survival of patients treated with this regimen.
* Determine the maximum percent reduction in tumor measurement in patients treated with this regimen.
* Collect blood and tissue from these patients for future correlative studies.

OUTLINE: This is an open-label, multicenter, dose-escalation study of erlotinib hydrochloride.

Patients receive oral sunitinib malate once daily on days 1-28 and oral erlotinib hydrochloride once daily on days 1-42. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 33% of patients experience dose-limiting toxicity. Once the MTD is determined, patients are treated with erlotinib hydrochloride at the MTD and sunitinib malate.

Patients undergo blood and tumor specimen collection periodically during study for future correlative studies.

PROJECTED ACCRUAL: A total of 49 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma with a component of clear cell or papillary carcinoma

  * Unresectable or metastatic disease (radiologically or clinically confirmed)
* Measurable disease (≥ 1 site)
* No known brain metastasis that has not been adequately treated with radiotherapy and/or surgery

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* No grade 3 hemorrhage within the past 4 weeks
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 times ULN (< 5 times ULN if due to underlying disease)
* No chronic liver disease (i.e., chronic active hepatitis or cirrhosis)
* Creatinine ≤ 1.5 times ULN
* None of the following cardiovascular conditions within the past 12 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
  * Ongoing cardiac dysrhythmia ≥ grade 2
  * Atrial fibrillation of any grade
  * Prolongation of the corrected QT (QTc) interval to > 450 msec for males or to > 470 msec for females
* Left Ventricular Ejection Fraction (LVEF) normal by Multigated Acquisition (MUGA) or echocardiogram
* No hypertension uncontrolled with medical therapy
* No other active malignancy within the past 5 years except basal cell skin cancer or cervical carcinoma in situ
* No uncontrolled adrenal insufficiency
* No uncontrolled hypothyroidism
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection)
* No impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior major surgery
* More than 4 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to > 25% of the bone marrow
* More than 28 days since prior investigational agents
* No prior sunitinib malate
* No prior anti-epidermal growth factor receptor therapy (e.g., erlotinib hydrochloride, panitumumab, cetuximab, or gefitinib)
* No concurrent therapeutic warfarin

  * Low-dose oral warfarin ≤ 2 mg daily for deep vein thrombosis prophylaxis is allowed after the maximum tolerated dose of erlotinib hydrochloride is determined
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent chemotherapy or biologic therapy
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2010-08 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. Ryan, MD, Study Chair — OHSU Knight Cancer Institute
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Salem Hospital, Salem, Oregon

REFERENCES:
- [Result] Ryan CW, Curti BD, Pattee KJ, et al.: A dose-escalation phase II study of sunitinib (S) plus erlotinib (E) in advanced renal carcinoma (RCC). [Abstract] American Society of Clinical Oncology 2008 Genitourinary Cancers Symposium, Feb 14-16, 2008, San Francisco, CA. A-361, 2008.
- [Derived] Feng Z, Curti BD, Quinn DI, Strother JM, Chen Z, Agnor R, Beer TM, Ryan CW. A Phase II, Single-arm Trial of Sunitinib and Erlotinib in Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2022 Oct;20(5):415-422. doi: 10.1016/j.clgc.2022.04.018. Epub 2022 May 5. PMID 35688679

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The discrepancy between the number of participants enrolled (60) and the number of participants Started in the Participant Flow module (46) is due to screen failures and consent withdrawals.
Groups:
- Sunitinib and Erlotinib: Erlotinib: Dose Level 0 = 50 mg/day, continuous daily; 0.5= 75 mg/day, continuous daily;
  1. 100 mg/day, continuous daily; 1.5= 125 mg/day, continuous daily;
  2. 150 mg/day, continuous daily
  Sunitinib: 50 mg daily, 4 weeks on, 2 weeks off
Period: Overall Study
Arm/Group | Sunitinib and Erlotinib
Started | 46
Completed | 43
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: The discrepancy between the number of participants enrolled (60) and the number of participants Started in the Participant Flow module (46) is due to screen failures and consent withdrawals.
Arm/Group | Sunitinib and Erlotinib
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 58 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Erlotinib Hydrochloride When Used in Combination With Sunitinib.
Description: The MTD is defined as the dose that produces dose limiting toxicity (DLT) in 33% of the patients.
Time Frame: Participants assessed for DLTs weekly during the first cycle of treatment and every 3 weeks in subsequent cycles until at least one DLT occurs in 33% or more of participants at that dose; participants assessed for the duration of the study, up to 7 years
Measure: Number; unit: milligrams
Arm/Group | Sunitinib and Erlotinib
Number analyzed (Participants) | 46
milligrams
  Sunitinib | 50
  Erlotinib | 150

2. Primary Outcome: Progression-free Survival at 8 Months
Description: Defined as the proportion of patients who are progression free (CR, PR and SD) at 8 months after initiating treatment with sunitinib in combination with erlotinib in patients with metastatic or unresectable clear cell or papillary carcinoma of the kidney. Complete Response (CR)= disappearance of all target lesions, Partial Response (PR)= At least a 30% decrease in the sum of the longest diameter of target lesions, and Stable Disease (SD)= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (20% increase in the sum).
Time Frame: 8 months after initiating treatment with sunitinib in combination with erlotinib in patients with metastatic or unresectable clear cell or papillary carcinoma of the kidney
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib and Erlotinib
Number analyzed (Participants) | 46
percentage of participants | 40 [23 to 56]

3. Secondary Outcome: To Determine the Safety of Sunitinib in Combination With Erlotinib
Time Frame: For the duration of the study, up to 7 years
Measure: Number; unit: participants
Arm/Group | Sunitinib and Erlotinib
Number analyzed (Participants) | 46
participants
  Diarrhea | 35
  Rash | 35
  Fatigue | 30
  Dysguesia | 29
  Nausea | 21
  Anorexia | 15
  Vomitting | 14
  Hand-foot syndrome | 13
  Stomatitis | 13
  Weight loss | 13
  Constipation | 12
  Dyspepsia | 12
  Dry skin | 10
  Alopecia | 9
  Pruritus | 9
  Other skin/hair changes | 8
  Dehydration | 5

4. Secondary Outcome: Median Time to Progression
Description: The Kaplan-Meier method will be used to estimate the median time to progression.
Time Frame: For the duration of the study, up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib and Erlotinib
Number analyzed (Participants) | 46
months | 5.8 [4.1 to 9.7]

5. Secondary Outcome: Proportion of Patients Whose Best Overall Response is Complete Response, Partial Response, Stable Disease, or Progressive Disease
Time Frame: From the start of treatment until the criteria for response is met.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib and Erlotinib
Number analyzed (Participants) | 46
percentage of participants
  Partial Response | 22
  Stable Disease | 59
  Progressive Disease | 11

6. Secondary Outcome: Maximum Percent Change in Tumor Measurement
Description: The maximum percent change in Tumor Measurement is the greatest percent change in longest diameter (LD) for the target lesions from the baseline LD. For patients with no change in LD, the maximum percent change is the lowest increase in LD from the baseline LD.
Time Frame: Baseline through end of study, up to 7 years
Measure: Mean (Full Range); unit: percent change in size
Arm/Group | Sunitinib and Erlotinib
Number analyzed (Participants) | 46
percent change in size | 18 [-100 to 94]

ADVERSE EVENTS:
Arm/Group | Sunitinib and Erlotinib
Serious Adverse Events (participants affected / at risk) | 7/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib and Erlotinib (N=46)
Hematuria (Renal and urinary disorders) | 1
Disease Progression (General disorders) | 1
Spontaneous Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Carcinoma of Prostatic Urethra (Renal and urinary disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 1
Abdominal Aortic Aneurysm (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib and Erlotinib (N=46)
Diarrhea (Gastrointestinal disorders) | 35
Rash (Skin and subcutaneous tissue disorders) | 35
Fatigue (General disorders) | 30
Dysguesia (Gastrointestinal disorders) | 29
Nausea (Gastrointestinal disorders) | 21
Anorexia (Gastrointestinal disorders) | 15
Vomitting (Gastrointestinal disorders) | 14
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 13
Stomatitis (Gastrointestinal disorders) | 13
Weight loss (General disorders) | 13
Constipation (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9
Other skin/hair changes (Skin and subcutaneous tissue disorders) | 8
Dehydration (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes